CLINICAL TRIAL: NCT00283101
Title: A Phase 1/2, Multi-Dose Study of SGN-40 (Anti-huCD40 mAb) in Patients With Chronic Lymphocytic Leukemia
Brief Title: A Safety Study in Patients With Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Seagen Inc. (Industry)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Jonathan Drachman, Sr. Medical Director, Seattle Genetics
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SG040-0003
Record Dates: First submitted 2006-01-25; First posted 2006-01-27 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2014-12

CONDITIONS: Leukemia, Lymphocytic, Chronic
Keywords: Antigens, CD40; Antibody, Monoclonal; Leukemia, Lymphocytic, Chronic, B-Cell; Hematologic Diseases; Immunoproliferatic Disorders; Lymphatic Diseases; Lymphoproliferative Disorders; Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Hematologic Diseases; Lymphatic Diseases; Lymphoproliferative Disorders; Leukemia | interventions — dacetuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): SGN-40
  Interventions: Drug: SGN-40 (anti-huCD40 mAb)

INTERVENTIONS:
Drug: SGN-40 (anti-huCD40 mAb) — 1-8 mg/kg IV; Days 1, 4, 8, 15, 22, 29 of Cycle 1 and Days 1, 15, 29 and 43 of Cycles 2-6.
  Other Names: dacetuzumab

SUMMARY:
This is an open-label, dose-escalation study to determine the tolerability, safety profile, and antitumor activity of SGN-40 in patients with CLL. All patients will receive dose escalation during the first two weeks regardless of cohort designation.

DETAILED DESCRIPTION:
A minimum of three patients will be entered into each dose-level cohort for five weeks. Escalation to the next cohort will occur when three patients have received at least one infusion at the highest scheduled dose level, and at least one patient has completed the entire five week dosing schedule. Cohorts will be enrolled at a maximal dose level of 3, 4, 6, or 8 mg/kg/week. Initial therapy will last for 5 weeks. Responding patients will receive additional infusions every two weeks x 4 at the maximal dose for each specific cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a histologic diagnosis of CLL as defined by the WHO criteria and exhibit active disease requiring treatment as per the NCI working group on CLL.
2. Patients must have a fresh tumor specimen available (peripheral blood or bone marrow) for flow cytometry evaluation (e.g. CD40, CD38, CD20, CD19, and CD5).For the phase 2 portion of the study, CD40 expression on malignant cells must be confirmed prior to registration.
3. Patients must have relapsed after receiving at least one fludarabine containing regimen or an equivalent purine analog.

   At study start patients must be at least 8 weeks or 5 plasma half-lives (whichever is greater) from prior chemotherapy/radiation/investigational agents, 8 weeks from prior antibody therapy and 6 months from autologous stem cell transplant.
4. Patients must have an ECOG performance status ≤ 2 and a life expectancy > 3 months.
5. Patients must have the following required baseline laboratory data:

   * Platelet count ≥ 50,000/mm3 (may be maintained by transfusion)
   * Hemoglobin ≥ 7.5 g/dL (may be maintained by transfusions or growth factors)
   * Absolute neutrophil count ≥ 1,000/mm3 (may be maintained by growth factors)
   * ALT/AST ≤ 2.0 times ULN
   * Total bilirubin ≤ 2.0 times ULN (unless related to hemolysis)
   * Creatinine < 2.0 times ULN
6. Females of childbearing potential must have a negative B-hCG pregnancy test result within 3 days prior to the first dose and must agree to use an effective contraceptive method during the course of the study and for 6 months following the last dose of study drug.
7. If a deep venous thrombosis or other vascular event has required medical or surgical intervention in the past year, patients must either: a) be on a stable dose of anticoagulant therapy (i.e., Coumadin and/or Heparin) for at least three weeks or b) have completed anticoagulant therapy at least three months prior to registration with radiographic confirmation that thrombosis is resolved. Prophylactic anticoagulant therapy for indwelling catheters is acceptable.
8. Patients must be at least 18 years of age.
9. Patients must be available for periodic blood sampling, study-related assessments, and management of toxicity at the treating institution.
10. Patients must give written informed consent. A copy of the signed informed consent form will be retained by the treating institution.

Exclusion Criteria:

1. Patients who have been treated previously with any anti-CD40 antibody.
2. Patients with a documented history within 6 months of registration of a cerebral vascular event (stroke or TIA), unstable angina, or myocardial infarction.
3. Patients with active CNS or leptomeningeal disease.
4. Patients who have received allogeneic stem cell transplant.
5. Patients who have had major surgery within four weeks prior to enrollment.
6. Patients with a known hypersensitivity to recombinant proteins or any excipient contained in the drug formulation.
7. Patients with a history of another primary malignancy that has not been in remission for at least 5 years (non-melanoma skin cancer and cervical carcinoma in situ on biopsy or a squamous intraepithelial lesion on PAP smear are exempt from the five year limit).
8. Patients with any systemic viral, bacterial, or fungal infection that has required antibiotic therapy within four weeks prior to enrollment. Prophylactic antibiotics and antiviral therapy are permitted prior to registration and are required during the study period (e.g. Bactrim, acyclovir).
9. Patients with known HIV, hepatitis B (by surface antigen expression), or active hepatitis C infection.
10. Patients on systemic steroids who have not been on a stable daily dose during the four weeks immediately prior to first dose of SGN-40. Maximum steroid dose is 10 mg prednisone per day or equivalent.
11. Patients with a history of migraines or severe headaches requiring medical therapy (other than occasional acetaminophen, aspirin, or non-steroidal anti-inflammatory drugs) within 12 months of enrollment.
12. Patients who are pregnant or breastfeeding.
13. Patients with any serious underlying medical condition that would impair their ability to receive or tolerate the planned treatment.
14. Patients with dementia or altered mental status that would preclude the understanding and/or rendering of informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2005-07; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD) of multiple doses of SGN-40
To evaluate the safety profile, immunogenicity, and pharmacokinetics of SGN-40
To test the antitumor activity of SGN-40 in patients with CLL who have demonstrated recurrence or progression after at least one systemic therapy

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Drachman, MD, Study Director — Seagen Inc.
Locations (4):
- United States (4):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Miami, Sylvester Comprehensive Cancer Center, Miami, Florida
  - Weill Medical College/Cornell University, New York, New York
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

REFERENCES:
- [Result] Furman RR, Forero-Torres A, Shustov A, Drachman JG. A phase I study of dacetuzumab (SGN-40, a humanized anti-CD40 monoclonal antibody) in patients with chronic lymphocytic leukemia. Leuk Lymphoma. 2010 Feb;51(2):228-35. doi: 10.3109/10428190903440946. PMID 20038235
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/20038235